CLINICAL TRIAL: NCT00321334
Title: Survival Study of Neo-adjuvant Versus Adjuvant Chemotherapy With Docetaxel Combined Carboplatin in Resectable Stage IB to IIIA Non-small Lung Cancer
Brief Title: Survival Study of Docetaxel and Carboplatin as Neo-Adjuvant Vs Adjuvant Chemotherapy in Early Stage NSLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese Society of Lung Cancer (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Professor, Chinese Society of Lung Cancer
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSLC0501
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; Chemotherapy; surgery; neo-adjuvant; adjuvant; RCT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetexel (Active Comparator): Chemotherapy+Surgery
  Interventions: Procedure: Chemotherapy+Surgery

INTERVENTIONS:
Procedure: Chemotherapy+Surgery — Docetaxel:75mg/m2 on D1 cycle,3 cycles Carboplatin:AUC=5 on D1 cycle,3 cycles

SUMMARY:
The objective of the trial is to determine whether 3 cycles of TP (docetaxel plus cisplatin) after complete operation will improve survival when compared with 3 cycles of TP prior to complete resection for NSCLC.

DETAILED DESCRIPTION:
Non-small-cell lung cancer (NSCLC) accounts for approximately 80% of lung cancers diagnosed worldwide. Surgical resection offers the best chance for cure for those patients diagnosed with early-stage disease, however, the vast majority of patients experience eventually relapse or metastasis. The rationale of neoadjuvant or adjuvant chemotherapy for early stage NSCLC lies in the possibility of eradicating micro-metastasis disease, so it appears to improve survival by reducing the occurrence of distant metastases. Meta analysis, CALGB 9633, JBR 10 and ANITA trials have shown postoperative (adjuvant) CT after complete resection will prolong survival. On the other hand, Depierre et al had conducted a trial to demonstrate preoperative (neoadjuvant ) chemotherapy in early stage NSCLC appears to improve survival. We need a head to head trial to comparing neoadjuvant with adjuvant chemotherapy to answer which treatment model is better to early stager NSCLC. Based on proven activity and survival benefit in advance NSCLC, docetaxel has been introduced into neoadjuvant therapy, even as a potential option in adjuvant setting.

Comparison: 3 cycles of TP after complete operation compared to 3 cycles of TP prior to complete resection for NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IB-IIIA non-small cell lung cancer patients,without previous chemotherapy, radiotherapy or target-therapy;
* age from 18 to 75;
* PS with ECOC 0-1;
* Adequate haematological and Hepatic- renal function;
* Expected to live longer than 12 months;
* The informed consent should be signed.

Exclusion Criteria:

* Patients with Small Cell Lung Cancer;
* Already receiving any prior anti-cancer treatment;
* Pregnant women;
* Uncontrolled diabetes, mental disease;
* Hepatic and renal function failure;
* The investigators believe the patient is not suitable to be enrolled in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2006-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
3 years Disease Free Survival (at end of 3 years) | Prospective

SECONDARY OUTCOMES:
3 years Overall Survival rate (at end of 3 years) and Safety data (after third cycle finish) | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long Wu, MD, FACS, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Chinese Society of Lung Cancer, Guangzhou, Guangdong, China